CLINICAL TRIAL: NCT05662059
Title: Investigating the Safety and Efficacy of Respiratory-Gated Auricular Vagal Afferent Nerve Stimulation (RAVANS) in Ulcerative Colitis (UC) in Pediatric and Young Adult Populations
Brief Title: Respiratory-gated Auricular Vagal Afferent Nerve Stimulation (RAVANS) Study in Ulcerative Colitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cala Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IBD-01
Record Dates: First submitted 2022-11-30; First posted 2022-12-22 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Sham-Controlled
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment (Experimental): Two therapy sessions (active stimulation) per day for 12 weeks with Treatment device
  Interventions: Device: RAVANS
- Sham (Sham Comparator): Two therapy sessions per day for 12 weeks with Sham device (no active stimulation)
  Interventions: Device: RAVANS-sham

INTERVENTIONS:
Device: RAVANS — Respiratory-Gated Auricular Vagal Afferent Nerve Stimulation
  Arms: Treatment
Device: RAVANS-sham — RAVANS sham device
  Arms: Sham

SUMMARY:
Prospective, single-center, sham-controlled, double-blinded 12-week study designed to evaluate the safety and efficacy of the RAVANS device in subjects with Ulcerative Colitis. The goal of the study is to distinguish sham (no stimulation) versus treatment (stimulation) response and to identify treatment responders. The study will last 12 weeks with in-clinic visits at 0 weeks and 12 weeks, and a telehealth-visit at week 6. Additionally, unscheduled visits may occur based on the needs of the subject or at the discretion of the investigator. Subjects will be randomized 2:1 to treatment or sham, and will stimulate at home twice per day.

ELIGIBILITY:
Inclusion Criteria:

1. Age 10-39 years
2. UC diagnosis for at least 3 months, confirmed by standard diagnostic evaluations including clinical, biochemical, and endoscopic studies
3. If age 17 years or younger, a PUCAI score of 10-60
4. A partial Mayo score of 3-6
5. If on corticosteroids, the dose must be stable and ≤ 10mg/day (prednisone or equivalent) for at least 14 days before entry into study
6. If on 5-Aminosalicylate, dose must be stable with following parameters:

   * 28 days on oral medication
   * 28 days on or off rectal medication
7. If on background immunosuppressive treatment the dose must be stable with the following parameters:

   * 56 days (8 weeks) for Immunomodulators (methotrexate, 6-MP, Azathioprine)
   * 112 days (16 weeks) for Infliximab, Adalimumab, Vedolizumab, Ustekinumab, other biologic, tofacitinib, upadacitinib, ozanimod
8. Able and willing to give written informed consent and comply with the requirements of the study protocol.
9. The earbud electrode must fit properly in the prospective subject's left ear
10. Fecal calprotectin of ≥150 during screening period

Exclusion Criteria:

1. Expectation to increase corticosteroids and/or immunosuppressive treatment
2. Presence of bowel stricture
3. History of intra-abdominal or perirectal abscess
4. Disease limited to only rectum (ulcerative proctitis)
5. Active treatment with antibiotics
6. Presence of active intestinal infection or documented infection by stool PCR or culture analysis in the previous 6 weeks
7. Continuous treatment with an anticholinergic medication, including over the counter medications (See appendix)
8. Implantable electronic devices such as pacemakers, defibrillators, hearing aids, cochlear implants or deep brain stimulators.
9. Current tobacco or nicotine user including nicotine patches, gum and vaping (to limit potential confounding effects of exposure to nicotine)
10. Bowel resection surgery within past 90 days prior to study enrollment, or planned surgery within the course of the study
11. Any planned surgical procedure requiring general anesthesia within the course of the study
12. Participation in any other Investigational drug and/or treatment currently or planned during the length of the study
13. Any condition which, in the opinion of the investigator, would jeopardize the subject's safety following exposure to a study intervention
14. Pregnancy or Lactation
15. Comorbid disease with high likelihood of requiring corticosteroid use
16. Inability to comply with study and follow-up procedures
17. Individuals with prior medical history of significant arrhythmias, including but not limited to, atrial fibrillation, atrial flutter, sick sinus syndrome, and AV blocks
18. Individuals with existing skin lesions on the left ear

Ages: 10 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Remission | 12 weeks
  Remission rate in treatment vs sham, assessed by a 0 or 1 point score in the Partial Mayo at week 12

SECONDARY OUTCOMES:
Clinical Responder | 12 weeks
  Responder rate in treatment vs sham, assessed by greater than or equal to a 2 point reduction in the Partial Mayo score at week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Feinstein Institute for Medical Research at Northwell Health, Lake Success, New York, United States